CLINICAL TRIAL: NCT05508282
Title: Reading Bees: Randomized Trial of an App-Based Approach to Reading (SHARE/STEP) and Screen Time Guidance for Parents of Infants During Pediatric Clinic Visits
Brief Title: Testing an App-Based Approach to Reading and Screen Time Guidance for Parents of Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: 2021-0635
Record Dates: First submitted 2022-02-22; First posted 2022-08-19 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Literacy; Parent-Child Relations; Language Development
MeSH Terms: conditions — Literacy

STUDY DESIGN:
Intervention Model Description: Single-blind randomized trial with two arms: intervention (enhanced reading & screen time guidance using a new mobile app) and control (usual guidance).
Who Masked: Participant
Masking Description: Parents will be advised of the purpose of the study in general terms (how parents and babies interact at home) yet not the behaviors or outcomes of interest.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): These parents will have a new mobile app (Reading Bees) installed onto their smartphone during a baseline clinic visit between 0 and 2-months old. They will also receive a specially designed children's book modeling the SHARE/STEP approach to reading with infants.
  At 6-months, these parents will also receive guidance regarding limiting digital media use (screen time) using content in the app and a specially designed children's book.
  They will also receive usual guidance during clinic visits via the Reach Out and Read program
  Interventions: Behavioral: Reading Bees app and children's book to enhance parent-infant reading quality (0-2 month visit); Behavioral: Reading Bees app and children's book to encourage alternatives to digital media (6-month visit)
- Control (No Intervention): These parents will receive usual reading and screen time guidance during pediatric clinic visits, including via the Reach Out and Read program.

INTERVENTIONS:
Behavioral: Reading Bees app and children's book to enhance parent-infant reading quality (0-2 month visit) — The reading intervention will be provided at the baseline clinic well-visit (0-2 months), and is based on the SHARE/STEP approach.
  Arms: Intervention
Behavioral: Reading Bees app and children's book to encourage alternatives to digital media (6-month visit) — The digital media (screen time) intervention will be provided at the 6-month clinic well-visit and is based on Baby Unplugged materials (book and app content).
  Arms: Intervention

SUMMARY:
The American Academy of Pediatrics (AAP) recommends that parents read to their children as often as possible beginning in infancy and limits on screen time at all ages, yet many families question the value of reading to infants and are uncertain how to do so, and screen time is rising. This proposal is highly relevant to public health in that it involves a "how-to" approach to reading with infants and limiting screen time that is delivered during pediatric well-child visits within an established program (Reach Out and Read) using innovative materials: specially designed children's books and animated educational videos featured in a new mobile app (Reading Bees). It addresses important research gaps, compliments existing programs and empowers families, particularly from underserved backgrounds, to read more interactively and enjoyably with their babies, limit screen time, and improve early literacy skills, relationships and health outcomes.

DETAILED DESCRIPTION:
The first year of life is a time of rapid brain development where critical skills, attitudes and routines predictive of academic, relational and health outcomes are shaped. An infant's home literacy environment (HLE), including quality of parent-child ("shared") reading, can be a major source of nurturing in these areas. Screen time in infancy can displace parent-child interaction and impair learning. The American Academy of Pediatrics (AAP) recommends shared reading from early infancy and discouraging screen time before 18-months old. While discussion of reading occurs in primary care, it is inconsistent and shared reading during infancy is modest. Screen time at this age is prevalent, increasing and hard to address. Reach Out and Read (ROR) provides books and guidance at well-visits from newborn to 5-years old and serves >5-million families/year. However, no structured approach to parent-infant reading has been developed. General urging to read at this age may be ineffective and fuel anxiety and "educational" screen time, especially in families of low-socioeconomic status (SES) with less experience. The long-term goal of this project is to establish a family-friendly approach to shared reading and screen time guidance in infancy. The objective of this application is to conduct a clinical trial of a "how-to" intervention alongside ROR compared to usual ROR, in families of low-SES. Intervention involves special children's books and videos in a new mobile app (Reading Bees). These introduce SHARE/STEP, a novel approach intended to enrich reading routines: Snuggle on lap, Hands on, show Affection, Respond (Stretch words, Talk about pictures, Explore sounds, Patience), Enjoy. A children's book encourages practice at home, and 3 animated videos provide extra guidance. Reading Bees also encourages parents to set goals, log daily reading and provides tips, awards and resources tailored to parent needs. Study staff will randomly enroll 93 families/group, collect Baseline data and deliver reading intervention at a Newborn, 1-month or 2-month visit. At the 6-month visit, screen time intervention will be introduced via the same approach (book, video in Reading Bees). Follow-up visits at 6- and 12-months will assess HLE, impression of materials, screen time and language. Reading and usage data will be accessed from Reading Bees app. Forty families/group will be invited to participate in video observation of shared reading in a private area prior to their child's 6- and 12-month old well-visit. These videos will be scored via two trained, independent coders applying both SHARE/STEP and social-emotional connection criteria (WECS scale). Our central hypothesis is that the Reading Bees intervention will be feasible during well-visits in early infancy, useful for families and effective to improve HLE and language and reduce screen time. The rationale is no similar intervention exists, current guidance is largely ineffective, and Reading Bees is synergistic and may be scaled within the ROR program and others such as home visiting. This research is significant and innovative in that it involves a novel approach to enhance parent-infant reading and limit screen time efficiently delivered during primary care, reinforces AAP guidelines and addresses NICHD/CDBB priority research areas. The expected outcome is successful testing of Reading Bees during a critical span of cognitive, relational and brain development, providing a foundation for further research and applications.

ELIGIBILITY:
Inclusion Criteria:

1. child age at enrollment less than 2.5 months old,
2. no documented history of neurologic insult, extreme prematurity (<32-weeks), or neurodevelopmental condition conveying risk of language delays,
3. custodial parent present is at least 18-years old,
4. custodial parent present is fluent in English without need of an interpreter, 5) child has no acute illness,
5. parent has an Android or iOS-compatible smartphone.

The subset of parent-child dyads recruited for video observation will be on a first-come, first-served basis from those enrolled in the parent study.

Exclusion Criteria:

Violating the above inclusion criteria.

Ages: 0 Months to 2 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 160 (Actual)
Dates: Start 2022-06-30 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Feasibility of intervention | Baseline visit (0-2 months)
  Feasibility of Reading Bees app for reading and screen time guidance; includes time of presentation and barriers encountered
Usability - reading and screen time materials | Baseline visit (0-2 months) for reading, 6-month visit for screen time. Higher scores suggest greater usability.
  Brief survey adapted from prior work involving anticipated usefulness and parental plans to use the infant reading book (SHARE This Book) and related content provided in the Reading Bees app. Items are categorical, Likert scale.
Efficacy - language | 12-month visit
  MacArthur-Bates Communicative Development Inventories, a validated parent-report measure of child language. Given time and possible literacy constraints, the Words & Gestures Short Form will be used.
Efficacy - change in quantitative home reading behaviors | Change between 6- and 12-month visits compared between groups.
  Books in the home, reading frequency and routines (StimQ Reading subscale). Higher score suggests more stimulating reading environment.
Efficacy - digital media use (screen time) | 12-month visit
  ScreenQ-I/T report measure/survey reflecting AAP screen time guidelines involving access to screens, frequency, content and co-viewing. Higher score reflects greater non-adherence with guidelines. Higher score suggests greater non-adherence with AAP guidelines and subsequently higher risk of adverse impacts. Range is 0-20 points.
Efficacy - change in qualitative home reading behaviors | Change between 6- and 12-month visits compared between groups.
  Shared reading quality/interactivity (SharePR report measure). Higher score suggests higher quality of shared reading. Range is 0-30 points.

SECONDARY OUTCOMES:
Video Observation of Shared Reading - Reading Quality | Change between 6- and 12-month visits compared between groups.
  A subset of parents (goal 40 per group) will be recruited for video observation of shared reading. Videos will be scored using a structured checklist of SHARE/STEP behaviors, with higher scores reflecting greater interactivity and reading quality.
Video Observation of Shared Reading - Change in Parent-Child Bonding | Change Between 6- and 12-month visits compared between groups.
  A subset of parents (goal 40 per group) will be recruited for video observation of shared reading. Videos will be scored using an established, observation-based measure of parent-child bonding (WECS), with higher scores reflecting greater connection.

CONTACTS AND LOCATIONS:
Overall Officials: John Hutton, MD, Principal Investigator — Assistant Professor
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2022-05-20): https://cdn.clinicaltrials.gov/large-docs/82/NCT05508282/ICF_000.pdf